CLINICAL TRIAL: NCT02747901
Title: Comparison Between Kinesiotaping and Cold Therapy on Muscle Strength and Functional Performance Outcomes After Total Knee Arthroplasty: a Randomized Controlled Trial
Brief Title: Comparison Between Kinesiotaping and Cold Therapy After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ertugrul Yuksel, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 1886-GOA
Record Dates: First submitted 2016-03-27; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Surgery
Keywords: KINESIOTAPING; COLD THERAPY; FUNCTIONAL PERFORMANCE
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Kinesiotaping Group (Experimental): Kinesiotaping group received kinesiotape for lymphatic correction and rectus femoris facilitation technique.
  Interventions: Other: KINESIOTAPING
- Cold Therapy Group (Active Comparator): Cold Therapy group received cold pack immediately after operation and following postoperative days.
  Interventions: Other: COLD THERAPY
- Control Group (No Intervention): Control group have no intervention.

INTERVENTIONS:
Other: KINESIOTAPING — Kinesiotaping group received kinesiotape for lymphatic correction and rectus femoris facilitation technique.
  Arms: Kinesiotaping Group
Other: COLD THERAPY — Cold therapy group received cold packs immediately after operation and following postoperative days
  Arms: Cold Therapy Group

SUMMARY:
The investigators aim was to compare the effectiveness of kinesiotaping and cold therapy on muscle strength and functional performance outcomes in patients with TKA during early postoperative period. One-hundred-eleven patents with TKA are going to randomly assigned to control, KT and CT groups (nC=nKT=nCT=37).

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) has been established as a valuable procedure patients with end-stage osteoarthritis and the rates of elective TKA are increasing steadily each year. Ninety percent of patients reported reduced pain, improved functional ability, and greater health related quality of life after TKA. Kinesiotaping (KT), a type of elastic tape that is being increasingly used for the management of pain and oedema after surgery

1. . Cold therapy (CT) can also help relieve pain and swelling during early postoperative period
2. . These two application may have impact on functional performance outcomes in patients with TKA. The number of studies that include KT in the rehabilitation process is increasing, but there isn't any study that compare KT application and CT after TKA.

The aim was to compare the effectiveness of kinesiotaping and cold therapy on muscle strength and functional performance outcomes in patients with TKA during early postoperative period.

Methods One-hundred-eleven patents with TKA are going to randomly assigned to control, KT and CT groups (nC=nKT=nCT=37). KT group are going to receive KT for lymphatic correction and rectus femoris facilitation technique. CT group are going to receive CT immediately after operation and following postoperative days. After surgery, all patients will receive standard post-operative treatment including continuous passive motion, active-assistive and active range of motion exercises, isometric and isotonic strengthening exercises, gait training and transfer training. After operation, pain intensity, active range of motion and knee function score [Hospital for Special Surgery (HSS) score] Functional activities are going to evaluate using the Iowa Level of Assistance Scale, and walking speed was evaluated using the Iowa Ambulation Velocity Scale. Isometric muscle strength measure of quadriceps femoris and hamstring muscles assessed by Hand-Held Dynamometer. All measurements evaluated at the discharge. One way ANOVA is going to be used in statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* 40 years older above
* have a primary total knee arthroplasty

Exclusion Criteria:

* revision total knee arthroplasty
* unable to understand verbal and written instructions
* having previously orthopaedic or neurological disorder that causes gait disturbance and having surgery within six months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
The maximum isometric muscle strength of Quadriceps and hamstring muscles of all the patients will be measured using Hand Held Dynamometer (Lafayette Instrument Company, Lafayette, Ind., USA). | Post-operative three months
  Before the measurement, the subjects seat with the hips on the edge of the bed, knees at ninety degree of flexion, feet free and arms crossed on the chest, without a support. The subjects complete maximum knee extension during the test. When the knee extension was achieved, the participant will be asked to continue maximum isometric contraction for five seconds. Then the mean value of three consecutive maximum contraction measurements will be taken. For the maximum isometric muscle strength of hamstring muscles of all the patients will be measured using Hand Held Dynamometer. Before the measurement, subjects lay prone on the bed, knees at ninety degree of flexion. Same measurement techniques will be used.

SECONDARY OUTCOMES:
Pain intensity of the knees will be measured by a numerical rating scale. | Post-operative three months
  Subjects will be asked to verbally rate the pain in and around the knee during activity and rest on the numeric rating scale from 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable.
The active knee range of motion will be measured using a full circle manual goniometer. | Post-operative three months
  The active knee range of motion will measured using a full circle manual goniometer made of flexible clear plastic with arms 30 cm in length. The patient will be positioned in the prone position.

CONTACTS AND LOCATIONS:
Overall Officials: Vasfi Karatosun, Prof, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, İ̇zmi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) are going to be kept.

REFERENCES:
- [Result] Donec V, Krisciunas A. The effectiveness of Kinesio Taping(R) after total knee replacement in early postoperative rehabilitation period. A randomized controlled trial. Eur J Phys Rehabil Med. 2014 Aug;50(4):363-71. Epub 2014 May 13. PMID 24819349
- [Result] Adie S, Kwan A, Naylor JM, Harris IA, Mittal R. Cryotherapy following total knee replacement. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD007911. doi: 10.1002/14651858.CD007911.pub2. PMID 22972114